CLINICAL TRIAL: NCT05036915
Title: The Effect of Routine and Random Pacifier Use Methods in Preterm Infants on Transition to Bottle Feeding Process
Brief Title: The Effect of Routine and Random Pacifier Use Methods in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Zehra Kan Onturk, Assist. Prof., Acibadem University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATADEK-2021/08
Record Dates: First submitted 2021-07-27; First posted 2021-09-08 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Feeding; Neonatal
Keywords: Preterm; Non-nutritive sucking; Feeding
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Pacifier randomly 30 min) (Experimental): Pacifier is randomly given to the infant for 30 min independent from feeding during the day
  Interventions: Procedure: Pacifier randomly
- Experimental Group (Pacifier randomly 30 min+ routine 5 min before each feeding) (Experimental): Pacifier is randomly given to the infant for 30 min independent from feeding during the day. In addition, pacifier is given to the infant for 5 min before each feeding.
  Interventions: Procedure: Pacifier other

INTERVENTIONS:
Procedure: Pacifier randomly — Common Action Steps:
  1. Legal representatives of newborns are informed about the study purpose, participants read and sign the informed consent form so their consent is obtained.
  2. Inclusion and exclusion criteria are evaluated.
  3. Study group is determined in line with the randomization order of the newborn to be included in the study.
  4. First part of the patient information and follow-up form is completed.
  5. Feeding content, amount and method are determined by the physician.
  Action Steps of the Control Group:
  * Pacifier is randomly given to the infant for 30 min independent from feeding during the day.
  1. Common procedure steps are applied.
  2. Procedure steps are applied in accordance with the "Neonatal Nursing Protocols" according to the newborn's feeding method.
  3. Second part of the patient information and follow-up form is completed daily.
  Arms: Control group (Pacifier randomly 30 min)
Procedure: Pacifier other — Procedure Steps of the Experimental Group:
  * Pacifier is randomly given to the infant for 30 min independent from feeding during the day. In addition, pacifier is given to the infant for 5 min before each feeding.
    1. Common procedure steps are applied.
    2. Pacifier is given for 5 min before each feeding.
    3. Procedure steps are applied in accordance with the "Neonatal Nursing Protocols" according to the newborn's feeding method.
    4. Second part of the patient information and follow-up form is completed daily.
  Arms: Experimental Group (Pacifier randomly 30 min+ routine 5 min before each feeding)

SUMMARY:
The aim of this study is to determine the effect of the routine 5-min pacifier use before feeding and the random 30-min pacifier use independent from feeding during the day on the transition to bottle feeding process in preterm infants.

DETAILED DESCRIPTION:
Preterm infants, may most frequently experience feeding difficulties as a result of lower oral-motor tone, poor coordination during sucking-swallowing-respiration, sleepy behavior, gastrointestinal dysmotility and immature sucking pressure and being unable to sustain their physiological values at a normal level during feeding. In the literature, it is reported that approximately 82% of preterm infants have an oral feeding difficulty. As a consequence, it is a very complex process to acquire a safe and effective feeding skill and preterm infants need support in the weeks after birth until participants develop skills that are necessary for oral feeding and complete a successful transition to total oral feeding independent from orogastric catheter.

Although studies have stressed positive effects of the Non-nutritive sucking (NNS) intervention on feeding performance, it is reported that there is a need for more comprehensive randomized controlled studies revealing the use frequency, duration or effect of time.

In the Neonatal Intensive Care Unit (NICU) where the study will be conducted, an appropriate method is chosen for preterm infants based on their general condition and the feeding transition stages are determined incrementally with repetitive follow-ups during feeding. The routine 5-min pacifier use method before feeding and the random 30-min pacifier use method during the day will be applied to newborns who have enteral feeding. Newborns who already use pacifier independent from feeding during the day in the clinic and to whom these methods are applied, will comprise the control group. In order to ensure a homogeneous application in the control group, the pacifier use duration will be limited to 30 minutes. Pacifier use durations have been determined in line with the literature examining the contribution of pacifier use to the feeding of preterm infants. Newborns, to whom the routine 5-min pacifier use method is applied before each feeding, will comprise the experimental group. All newborns included in the study will be followed until participants are discharged.

ELIGIBILITY:
Inclusion Criteria:

Preterm infants;

* Whose legal representatives agree to take part in the study and sign the informed consent form,
* Who have a stable clinical picture,
* Who are on the first day of enteral feeding will be included in the study.

Exclusion Criteria:

Preterm infants;

* Who have a comorbidity,
* Who are intubated,
* Who have an inherent anomaly,
* Who have parenteral feeding will not be included in the study.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Change in feed intake | From baseline to transition to total oral feeding (average 15 weeks)
  Change in feed intake will be assessed from baseline to transition to total oral feeding
Change in body weight | From baseline to transition to total oral feeding (average15 weeks)
  Participant's body weight will be assessed from baseline to transition to total oral feeding up to through study completion
Length of hospital stay | From baseline to discharge (average 15 weeks)
  The time from date of hospitalization until the date of discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Kan Öntürk, Assist Prof, Principal Investigator — Acibadem University
Locations (1):
- Acıbadem University Atakent Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dur S, Gozen D. Nonnutritive Sucking Before Oral Feeding of Preterm Infants in Turkey: A Randomized Controlled Study. J Pediatr Nurs. 2021 May-Jun;58:e37-e43. doi: 10.1016/j.pedn.2020.12.008. Epub 2021 Jan 6. PMID 33422394
- [Result] Foster JP, Psaila K, Patterson T. Non-nutritive sucking for increasing physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2016 Oct 4;10(10):CD001071. doi: 10.1002/14651858.CD001071.pub3. PMID 27699765
- [Result] Fucile S, Phillips S, Bishop K, Jackson M, Yuzdepski T, Dow K. Identification of a Pivotal Period in the Oral Feeding Progression of Preterm Infants. Am J Perinatol. 2019 Apr;36(5):530-536. doi: 10.1055/s-0038-1669947. Epub 2018 Sep 12. PMID 30208500
- [Result] Ostadi M, Jokar F, Armanian AM, Namnabati M, Kazemi Y, Poorjavad M. The effects of swallowing exercise and non-nutritive sucking exercise on oral feeding readiness in preterm infants: A randomized controlled trial. Int J Pediatr Otorhinolaryngol. 2021 Mar;142:110602. doi: 10.1016/j.ijporl.2020.110602. Epub 2020 Dec 29. PMID 33412344
- [Result] Pineda R, Dewey K, Jacobsen A, Smith J. Non-Nutritive Sucking in the Preterm Infant. Am J Perinatol. 2019 Feb;36(3):268-276. doi: 10.1055/s-0038-1667289. Epub 2018 Aug 6. PMID 30081403